CLINICAL TRIAL: NCT03571269
Title: Effective ReperfusiOn Strategy for Patients With ST-segment Elevation Myocardial Infarction Guided by Optical Coherence Tomography Versus ANgiography (EROSION III): a Multicenter, Randomized Controlled Trial
Brief Title: EROSION III: OCT- vs Angio-based Reperfusion Strategy for STEMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harbin Medical University (Other)
Collaborators: Second Hospital of Jilin University (Other); Daqing Oil Field Hospital (Other); Tianjin Chest Hospital (Other); Second Affiliated Hospital of Nanchang University (Other); First Affiliated Hospital of Xinjiang Medical University (Other); Beijing Anzhen Hospital (Other); First Affiliated Hospital of Guangxi Medical University (Other); Peking University First Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); The Second Hospital of Hebei Medical University (Other); The Second Affiliated Hospital of Dalian Medical University (Other)
Responsible Party: Principal Investigator, Yu Bo, Director, Harbin Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016YFC1301103
Record Dates: First submitted 2018-06-15; First posted 2018-06-27 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: ST-segment Elevation Myocardial Infarction
Keywords: STEMI; optical coherence tomography; reperfusion
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OCT-guided group (Experimental): Detailed methods of OCT examination are the same as above. Whether stenting or not will be decided by the operators according to the underlying mechanisms of culprit lesions. If stenting, OCT will be used to guide and optimize the whole process of PCI. Patients will be treated with dual antiplatelet therapy (aspirin+ticagrelor or aspirin+clopidogrel) for at least 12 months.
  Interventions: Procedure: Optical coherence tomography-guided reperfusion strategy
- Angiography-guided group (No Intervention): Detailed methods of angiography examination are the same as above. Whether stenting or not and the whole process of PCI will be decided by the operators according to the current treatment standard of angiography. Patients will be treated with dual antiplatelet therapy (aspirin+ticagrelor or aspirin+clopidogrel) for at least 12 months.

INTERVENTIONS:
Procedure: Optical coherence tomography-guided reperfusion strategy — Optical coherence tomography will be used to detect the detailed characteristics of culprit lesion and to decide and optimize the reperfusion strategy according to the established algorithm in the protocol.
  Arms: OCT-guided group

SUMMARY:
Brief Summary: This study is a prospective, multicenter, randomized, controlled trial aimed to compare the reperfusion strategy and clinical outcomes of STEMI patients treated by angiography-guided vs. OCT-guided PCI. Patients presenting STEMI with coronary artery diameter stenosis ≤70% and TIMI blood flow grade 3 at index or after thrombus aspiration are randomly assigned to either an OCT-guided group or an angiography-guided group. In OCT-guided group, stent implantation or conservative medical treatment is determined based on OCT findings. Conservative non-stenting strategy will be recommended in those with culprit plaque erosions, certain ruptures without dissection and hematoma, SCAD without obstructive stenosis. In the angiography-guided group, reperfusion strategy is decided by the operators according to the local practice. The rate of stenting during primary PCI and clinical outcomes at 1-month and 1-year are collected.

DETAILED DESCRIPTION:
Methodology: As a multicenter, prospective, randomized, controlled trial, patients with ST-segment elevation myocardial infarction (STEMI) who have an intermediate stenotic culprit lesion (angiographic diameter stenosis ≤70%) and TIMI flow grade 3 or residual stenosis ≤70% after thrombus aspiration and TIMI grade 3 will be enrolled and randomized to OCT-guided group or angiography-guided group. In OCT-guided group, pre-PCI OCT imaging of the culprit lesion will be performed and revascularization strategy will be determined based on underlying mechanism of culprit lesion morphology. For lesions required stenting, OCT measurements will be used to guide the selection of stent size and to optimize the result of stent implantation. In the angiography-guided group, OCT will not be performed and the PCI procedures will be done according to routine practice by the operators. Primary outcome is patient-level rate of stenting during primary PCI and the incidence of recurrent myocardial ischemic events (unstable angina-induced rehospitalization, recurrent myocardial infarction, target lesion revascularization) or cardiac death within 1 month. Secondary outcomes include the incidence of cardiocerebrovascular events (cardiac death, recurrent myocardial infarction, stroke, target lesion revascularization, malignant arrhythmia, and unstable angina-induced rehospitalization) and the incidence of heart failure event within 1 year.

Patient enrollment and procedure overview: Patients with STEMI<12h in whom coronary angiography is planned will be screened. Those have a culprit lesion stenosis ≤70% by visual estimation and TIMI blood flow grade 3 at index angiography or after thrombus aspiration will be consented to participate in the study. After informed consent obtained, patients will be assigned to OCT-guided group or angiography-guided group randomly. In the OCT-guided group, OCT imaging of infarcted-related artery will be performed to assess the underlying mechanism of culprit lesion. Reperfusion strategy will be decided by the operators according to the OCT findings. Conservative medical strategy will be recommended if the underlying mechanism is plaque erosions, small ruptures without dissection and hematoma, SCAD without obstructive stenosis. Otherwise, stent implantation may be performed. The procedure of stent implantation will be guided by OCT according to current guideline and consensus documents. Before stent implantation, the landing zone and size of stent will be decided according to the pre-PCI OCT images. After implantation, OCT imaging will be performed to optimize the results of stent implantation including stent expansion, apposition, edge dissection, tissue protrusion. In the angiography-guided group, PCI procedure will be performed according to current guidelines and their daily practice. All patients are required to take dual antiplatelet treatment with aspirin (100 mg/day) and ticagrelor (180 mg/day) or clopidogrel (75mg/day) for at least 12 months. The use of low molecular weight heparin and glycoprotein IIb/IIIa inhibitor are determined by the operators.

Follow-up: Patients will be followed by phone calls or clinical visits by study coordinators at 1 month (30 days) and 1 year (12 months). Severe adverse events including heart failure event, stent failure, cardiac death, recurrent myocardial infarction, stroke, target lesion revascularization, malignant arrhythmia, and unstable angina-induced rehospitalization will be collected in all patients throughout the whole study period until the last patient completes 12 months of follow up. Additional phone follow-up may also be performed subject to executive committee approval.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old ≤ age ≤ 80 years old;
2. Patients with STEMI<12h;
3. The target lesion is located in a native coronary artery;
4. The residual diameter stenosis (DS) is ≤70% on angiogram and thrombolysis in myocardial infarction (TIMI) flow grade is 3 after thrombus aspiration or not;
5. Written informed consent.

Exclusion Criteria:

1. Patients who are breastfeeding or pregnant or planning to pregnant during the study period;
2. Patients with a history of heart failure;
3. Hemodynamic instability;
4. Target lesion such as: left main coronary artery; three-vessel disease; ostial lesion (defined as within 3mm of the left main coronary artery or aorto-ostium); tortuous lesion; angular lesion;
5. Subjects with contraindication of contrast medium;
6. There are contraindications to aspirin or clopidogrel;
7. Severe hepatic and renal insufficiency (ALT or AST >3x upper limits of normal, creatinine>2.0 mg/dL or end-stage renal disease);
8. Patients with bleeding tendency such as peptic ulcer, bleeding or coagulation disorders;
9. AMI is caused by surgery, trauma, gastrointestinal bleeding, PCI, or its complications;
10. AMI occurs in patients who have been hospitalized for other reasons;
11. Patients who were considered with poor compliance and could not complete the study as required judged by the investigators;
12. Patient with life expectancy ≤24 months;
13. Patients with heart transplantation;
14. Patients with definite diagnosis of tumors;
15. Patients who are currently enrolled in other clinical trial (except other subjects in this project) which has not reached its primary endpoint;
16. Patients who are not suitable for the current study judged by the investigators.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2020-01-02 (Actual); Study Completion 2020-12-24 (Actual)

PRIMARY OUTCOMES:
Primary effective endpoint of OCT-guided reperfusion strategy (powered) | Immediate after primary PCI
  Patient-level rate of stent implantation between the two groups
Primary safety endpoint of OCT-guided reperfusion strategy | Within 1 month
  The incidence of recurrent myocardial ischemic events (unstable angina-induced rehospitalization, recurrent myocardial infarction, target lesion revascularization) or cardiac death.

SECONDARY OUTCOMES:
Incidence of cardiocerebrovascular events | Within 1 year
  Cardiocerebrovascular events include cardiac death, recurrent myocardial infarction, stroke, target lesion revascularization, malignant arrhythmia, and unstable angina-induced rehospitalization.
Incidence of heart failure event | Within 1 year
  Heart failure is a complex syndrome in which ventricular filling or ejection fraction is impaired due to structural or functional abnormality of the heart.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Yu, Study Chair — The Second Affiliated Hospital of Harbin Medical University; Bin Liu, Principal Investigator — Second Hospital of Jilin University; Jianping Li, Principal Investigator — Peking University First Hospital; Yanqing Wu, Principal Investigator — Second Affiliated Hospital of Nanchang University; Ling Li, Principal Investigator — The First Affiliated Hospital of Zhengzhou University; Chunmei Wang, Principal Investigator — Beijing Anzhen Hospital; Yin Liu, Principal Investigator — Tianjin Chest Hospital; Dajun Yuan, Principal Investigator — The Second Affilated Hospital of Dalian Medical University; Zhiqi Sun, Principal Investigator — Daqing Oil Field Hospital; Yining Yang, Principal Investigator — First Affiliated Hospital of Xinjiang Medical University; Xinshun Gu, Principal Investigator — The Second Hospital of Hebei Medical University; Lang Li, Principal Investigator — First Affiliated Hospital of Guangxi Medical University
Locations (12):
- China (12):
  - Beijing Anzhen Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Daqing Oil Field Hospital, Daqing, Heilongjiang
  - The 2nd Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Second Hospital of Jilin University, Jilin, Jilin
  - The Second Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality
  - First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang

REFERENCES:
- [Derived] Jia H, Dai J, He L, Xu Y, Shi Y, Zhao L, Sun Z, Liu Y, Weng Z, Feng X, Zhang D, Chen T, Zhang X, Li L, Xu Y, Wu Y, Yang Y, Wang C, Li L, Li J, Hou J, Liu B, Mintz GS, Yu B. EROSION III: A Multicenter RCT of OCT-Guided Reperfusion in STEMI With Early Infarct Artery Patency. JACC Cardiovasc Interv. 2022 Apr 25;15(8):846-856. doi: 10.1016/j.jcin.2022.01.298. Epub 2022 Mar 30. PMID 35367176